CLINICAL TRIAL: NCT06374043
Title: Individual Albuminuria Lowering Response to Dapagliflozin in a Decentralized Clinical Trial in Patients With Type 2 Diabetes Mellitus and Elevated Albuminuria
Brief Title: Decentralized N=1 Study: A Feasible Approach to Evaluate Individual Therapy Response to Dapagliflozin.
Acronym: @HOME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/1002
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus Type 2 With Proteinuria; Diabetes Mellitus; Diabetes; Diabetes Complications; Albuminuria; Chronic Kidney Diseases; Chronic Kidney Disease Due to Type 2 Diabetes Mellitus; CKD; Proteinuria
Keywords: Type 2 diabetes; Diabetes Mellitus, Type 2; Albuminuria; Diabetes Mellitus; Diabetes Mellitus Type 2 with Proteinuria; Personalized Medicine; Decentralized; Remote clinical trial; Remote data collection; Individualized; CKD; Chronic Kidney Disease; Albuminuria-Lowering therapies; Dapagliflozin; SGLT2 inhibitor; Placebo-controlled; Randomized; Cross-over; N=1; N-1; Sodium Glucose Co-Transporter 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetes Complications; Albuminuria; Renal Insufficiency, Chronic; Proteinuria | interventions — dapagliflozin; Micro-Electrical-Mechanical Systems

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind cross-over trial with repeated administration (i.e., a series of N=1 trials).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Option 1 (D-D-P-P) (Other): Week 1. Dapagliflozin 10 mg/day Week 2. Wash-out Week 3. Dapagliflozin 10 mg/day Week 4. Wash-out Week 5. Placebo Week 6. Wash-out Week 7. Placebo Week 8. Wash-out
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Placebo; Device: Withings BPM Connect; Device: Withings Body+; Diagnostic Test: Hem-Col Capillary Blood Collection Device; Device: MEMS (Medication Electronic Monitoring System) Cap; Behavioral: Questionnaire: participants' perspectives toward remote data collection
- Option 2 (D-P-D-P) (Other): Week 1. Dapagliflozin 10 mg/day Week 2. Wash-out Week 3. Placebo Week 4. Wash-out Week 5. Dapagliflozin 10 mg/day Week 6. Wash-out Week 7. Placebo Week 8. Wash-out
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Placebo; Device: Withings BPM Connect; Device: Withings Body+; Diagnostic Test: Hem-Col Capillary Blood Collection Device; Device: MEMS (Medication Electronic Monitoring System) Cap; Behavioral: Questionnaire: participants' perspectives toward remote data collection
- Option 3 (D-P-P-D) (Other): Week 1. Dapagliflozin 10 mg/day Week 2. Wash-out Week 3. Placebo Week 4. Wash-out Week 5. Placebo Week 6. Wash-out Week 7. Dapagliflozin 10 mg/day Week 8. Wash-out
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Placebo; Device: Withings BPM Connect; Device: Withings Body+; Diagnostic Test: Hem-Col Capillary Blood Collection Device; Device: MEMS (Medication Electronic Monitoring System) Cap; Behavioral: Questionnaire: participants' perspectives toward remote data collection
- Option 4 (P-P-D-D) (Other): Week 1. Placebo Week 2. Wash-out Week 3. Placebo Week 4. Wash-out Week 5. Dapagliflozin 10 mg/day Week 6. Wash-out Week 7. Dapagliflozin 10 mg/day Week 8. Wash-out
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Placebo; Device: Withings BPM Connect; Device: Withings Body+; Diagnostic Test: Hem-Col Capillary Blood Collection Device; Device: MEMS (Medication Electronic Monitoring System) Cap; Behavioral: Questionnaire: participants' perspectives toward remote data collection
- Option 5 (P-D-P-D) (Other): Week 1. Placebo Week 2. Wash-out Week 3. Dapagliflozin 10 mg/day Week 4. Wash-out Week 5. Placebo Week 6. Wash-out Week 7. Dapagliflozin 10 mg/day Week 8. Wash-out
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Placebo; Device: Withings BPM Connect; Device: Withings Body+; Diagnostic Test: Hem-Col Capillary Blood Collection Device; Device: MEMS (Medication Electronic Monitoring System) Cap; Behavioral: Questionnaire: participants' perspectives toward remote data collection
- Option 6 (P-D-D-P) (Other): Week 1. Placebo Week 2. Wash-out Week 3. Dapagliflozin 10 mg/day Week 4. Wash-out Week 5. Dapagliflozin 10 mg/day Week 6. Wash-out Week 7. Placebo Week 8. Wash-out
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Placebo; Device: Withings BPM Connect; Device: Withings Body+; Diagnostic Test: Hem-Col Capillary Blood Collection Device; Device: MEMS (Medication Electronic Monitoring System) Cap; Behavioral: Questionnaire: participants' perspectives toward remote data collection

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Oral administration
  Other Names: Forxiga; (2S,3R,4R,5S,6R)-2-[4-chloro-3-(4-ethoxybenzyl)phenyl]-6-(hydroxymethyl)tetrahydro-2H-pyran-3,4,5-triol; A10BK01
Drug: Placebo — Oral administration
Device: Withings BPM Connect — CE marked and clinically validated blood pressure monitor. Clinical trial results are within the margin of acceptance defined by the internationally recognized evaluation standard of blood pressure monitors ANSI/AAMI/ISO 81060-2:2013, EN ISO 81060-2:2014, developed by the European Society of Hypertension, British Hypertension Society and Association for the Advancement of Medical Instrumentation/American Heart Association.
  Blood pressure will be measured by the participants once daily on 28 days. Three consecutive measurements are taken.
Device: Withings Body+ — CE marked and clinically validated advanced Wi-Fi smart scale.
  Body weight will be measured by the participants once daily on 40 days.
Diagnostic Test: Hem-Col Capillary Blood Collection Device — Capillary blood samples will be obtained using a BD Microtainer® Contact-Activated Lancet (Franklin Lakes, New Jersey, USA) once daily on 22 days. These blood samples will be collected into Hem-Col® tubes (Hem-Col, Labonovum, Limmen, the Netherlands), specifically designed for collection of capillary blood acquired through a finger prick. The Hem-Col microtube is equipped with an anticoagulant and a preservation buffer, enhancing the stability of analytes in whole blood. These Hem-Col tubes have the dimensions of standard blood collection tubes and are constructed from polyethylene, featuring a pierceable cap made of thermoplastic elastomers. Each tube incorporates a liquid barrier, with the inner part preventing the loss of Hem-Col preservation fluid and the outer part serving as a scoop for collecting blood from a finger prick. The Hem-Col lithium heparin tubes will be utilized for the analysis of creatinine, CRP, lipid profile, HbA1c, uric acid, glucose and NT-proBNP.
Device: MEMS (Medication Electronic Monitoring System) Cap — Medication will be provided in standard medicine bottles with the MEMS® (Medication Electronic Monitoring System) Cap (AARDEX Ltd, Union City, CA, USA), which is a customizable medication package which records and stores up to 4,000 dosing events. The cap fits on standard medicine bottles and with integrated microcircuits, the child-resistant MEMS® Cap records the date and time whenever a patient opens a vial. The stored information can be transferred at any time through the MEMS® Reader to the adherence software for immediate analysis and interpretation.
Behavioral: Questionnaire: participants' perspectives toward remote data collection — Self-made questionnaires consisting of 6 multiple choice questions and 2 open questions will be used to assess patient experience and satisfaction to guide and inform future trials and use in clinical practice.

SUMMARY:
Randomized placebo-controlled double-blind cross-over N=1 trial in adult male and female patients with UACR >20 mg/g (2.26 mg/mmol) with type 2 diabetes treated in primary or secondary healthcare.

The goal of this clinical trial is to determine the individual response to the SGLT2 inhibitor dapagliflozin in urine albumin-to-creatinine ratio (UACR). Secondary objectives are to determine the individual response to dapagliflozin in systolic blood pressure, body weight, eGFR, and fasting plasma glucose.

Participants will collect all study data in the comfort of their own environments:

* First-morning void urine samples
* Capillary blood samples
* Blood pressure
* Body weight

Participants will be randomly assigned to a cross-over study consisting of two periods of 1-week treatment with dapagliflozin 10 mg/day and two periods of 1-week treatment with placebo in random order with a 1-week wash-out period between every treatment period to avoid cross-over effects.

DETAILED DESCRIPTION:
Rationale:

Persistent increased albuminuria is a strong risk marker for progressive kidney disease and cardiovascular disease in patients with or without diabetes. The degree of albuminuria reduction in the first months of treatment with pharmacological or dietary intervention correlates with the degree of long-term (3 to 4 years) renal or cardiovascular protection. Despite the various available treatments to decrease urinary albumin excretion, residual albuminuria persists in many patients. The high residual albuminuria in a proportion of patients is at least in part explained by suboptimal response to the current treatments (i.e., ACE inhibitor or Angiotensin Receptor Blockers).

Dapagliflozin is a sodium-glucose transport inhibitor and inhibits the reabsorption of glucose in the proximal tubule. This leads to a decrease in fasting plasma glucose and HbA1c in patients with type 2 diabetes. In addition, dapagliflozin administration causes a decrease in blood pressure and body weight and an increase in hematocrit suggestive of a diuretic effect. Previous studies have also demonstrated the albuminuria lowering effects of dapagliflozin in patients with type 2 diabetes mellitus.

Although dapagliflozin markedly slows progression of kidney function decline (and reduces cardiovascular outcomes) on a population level, randomized parallel group trials have suggested a marked variation in the response to dapagliflozin between individual patients. By design, randomized parallel group placebo-controlled clinical trials test the efficacy of new interventions on a population level but do not assess the efficacy of a drug for the individual. Although there is variation in response between patients, parallel group trial does not allow conclusions whether this variation is a true variation in drug response, or measurement or temporal random variation. The investigators therefore propose a cross-over trial with repeated administration (i.e., a series of N=1 trials) to ascertain the individual drug response. This design specifically allows for assessment of drug efficacy and safety at an individual level.

Objectives:

* Primary: To determine the individual response to the SGTL2 inhibitor dapagliflozin in urine albumin-to-creatinine ratio (UACR)
* Secondary: To determine the individual response to the SGLT2 inhibitor dapagliflozin in: systolic blood pressure, body weight, eGFR, fasting plasma glucose

Study design:

Randomized placebo-controlled double-blind cross-over N=1 trial. Eligible participants will be invited for screening. After a screening visit, eligible patients will be randomly assigned to a cross-over study consisting of two periods of 1-week treatment with dapagliflozin and two periods of 1-week treatment with placebo in random order with a 1-week wash-out period between every treatment period to avoid cross-over effects. Based on a prior study where patients were exposed to dapagliflozin 10 mg, effects of dapagliflozin on UACR, blood pressure, body weight, eGFR and plasma glucose were fully present after 1 week and returned to baseline 4 days after drug discontinuation. Hence, a 1-week treatment followed by 1 week wash-out is considered sufficient to detect treatment effects.

Study population:

Adult male and female patients with UACR >20 mg/g (2.26 mg/mmol) with type 2 diabetes mellitus treated in primary or secondary healthcare. Subjects will be recruited via general practitioner practices and via the outpatient clinic of the Department of Internal Medicine of the Ziekenhuisgroep Twente, Almelo.

Intervention:

Dapagliflozin 10 mg/day

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The efficacy and safety of dapagliflozin is established in multiple parallel randomized controlled trials involving more than 25,000 patients with type 2 diabetes. Urinary tract infections and genital infections are the most frequently reported side effects. Dapagliflozin reduces body weight unlike sulfonylurea derivatives and insulin.

Participants visit the outpatient clinic at three occasions (i.e., a screening visit, a second visit and end of study visit) and have to record body weight and blood pressure at home and collect blood and urine at home.

Blood pressure and body weight are measured at home by the participants using ambulant devices (Withings BPM Connect and Withings Body+, respectively). Participants measure their blood pressure and body weight once daily on 28 and 40 days in total, respectively. Capillary blood will be sampled at home by participants using a BD Microtainer® Contact-Activated Lancet (once daily on 22 days in total). Blood is collected with the Hem-Col® device, which is designed to collect capillary blood drawn with a finger prick. In order to make patients comfortable with the blood collection procedures, they first collect a capillary blood sample at the study site during the second visit under supervision of trained lab technicians. A venous blood sample will also be taken during the second visit in order to compare the clinical chemistry assessments in capillary blood with those measured in venous blood samples (NL70447.100.19). Participants will be asked to draw blood samples at home by a finger prick and send the samples to the laboratory. Participants will collect first morning void urine samples through the PeeSpot® device (once daily on 40 days in total) which allows for decentralized urine collection in a small tube. The urine tubes and blood samples will be sent by regular mail to the laboratory. No other invasive measurements will be executed.

The advantage of an N=1 study is that efficacy of the intervention is vetted for the actual participant. Dapagliflozin is currently marketed in the Netherlands and recommended in patients with type 2 diabetes mellitus and eGFR>45 mL/min/1.73m2. Patients who show a satisfactory response to dapagliflozin and whose characteristics fulfill the criteria according to which dapagliflozin can be prescribed in clinical practice are offered to receive dapagliflozin after the study. It is expected that the indication for dapagliflozin will be broadened to patients with eGFR 25-45 mL/min/1.73m2 in the near future. If this occurs, these patients can also be treated on-label in practice.

The expected time investment for participants is 20 hours, including measurements at home. Participants receive restitution of travel costs to visit the outpatient clinic for the screening, randomization and end of study visit. Participants receive no priority in treatment of other diseases in the clinic during this study. Participation in this study is on a free-will base. Participants can keep the body weight scale and blood pressure device at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of type 2 diabetes mellitus
* Urinary albumin-to-creatinine ratio >20 mg/g (2.26 mg/mmol)
* eGFR >30 ml/min/1.73m2
* Willing to sign informed consent

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Prior treatment with SGLT2 inhibitor in the four weeks prior to randomization
* History of severe hypersensitivity or contraindications to dapagliflozin
* Unable to monitor blood pressure / body weight or handle digital technologies
* History of non-adherence to medical regimens or unwillingness to comply with the study protocol
* Participation in any clinical investigation within 3 months prior to initial dosing
* Unstable or rapidly progressing renal disease
* Severe hepatic impairment (Child-Pugh class C) as determined by the treating physician.
* Active malignancy
* Any medication, surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of medications including, but not limited to any of the following: History of active inflammatory bowel disease, within the last six months; Major gastrointestinal tract surgery as decided by the treating physician; Pancreatitis within the last six months; Evidence of serious hepatic disease as determined by the treating physician; Evidence of urinary obstruction or difficulty in voiding at screening.
* Confirmed lactose intolerance demonstrated with a lactose intolerance test.
* Donation or loss of 400 mL of blood within 8 weeks prior to initial dosing
* History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during the screening
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* Current pregnancy or breast feeding / attempting to conceive.
* Women of childbearing potential (WOCBP): WOCBP who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of study drug in such a manner the risk of pregnancy is minimized; WOCBP must have a negative serum or urine pregnancy test result (minimum sensitivity 25 IU/L or equivalent of HCG) within 0 to 72 hours before the first dose of study drug.

WOCBP comprises women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who are not post-menopausal (see definition below). The following women are WOCBP:

* Women using the following methods to prevent pregnancy: oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as intrauterine devices or barrier methods (diaphragm, condoms, spermicides).
* Women who are practicing abstinence.
* Women who have a partner who is sterile (e.g. due to vasectomy).

Post-menopause is defined as:

* Women who have had amenorrhea for >12 consecutive months (without another cause) and who have a documented serum follicle-stimulating hormone (FSH) level >35 mIU/mL.
* Women who have irregular menstrual periods and a documented serum FSH level >35 mIU/mL.
* Women who are taking hormone replacement therapy (HRT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
UACR response | Will be assessed within 6 months and reported within 1.5 years after conclusion of the study.
  The individual response to the SGLT2 inhibitor dapagliflozin in urine albumin-to-creatinine ratio (UACR)

SECONDARY OUTCOMES:
Systolic blood pressure response | Will be assessed within 6 months and reported within 1.5 years after conclusion of the study.
  The individual response to the SGLT2 inhibitor dapagliflozin in systolic blood pressure.
Body weight response | Will be assessed within 6 months and reported within 1.5 years after conclusion of the study.
  The individual response to the SGLT2 inhibitor dapagliflozin in body weight.
eGFR response | Will be assessed within 6 months and reported within 1.5 years after conclusion of the study.
  The individual response to the SGLT2 inhibitor dapagliflozin in eGFR.
Fasting plasma glucose response | Will be assessed within 6 months and reported within 2 years after conclusion of the study.
  The individual response to the SGLT2 inhibitor dapagliflozin in glucose.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Ziekenhuisgroep Twente, Almelo
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Yes